CLINICAL TRIAL: NCT00165178
Title: Treatment of Acute Lymphoblastic Leukemia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Children's Hospital (Other); University of Rochester (Other); McMaster University (Other); San Jorge Children's Hospital (Puerto Rico) (Unknown); St. Justine's Hospital (Other); Maine Children's Cancer Program (Other); Ochsner Health System (Other); Tulane University School of Medicine (Other); Laval University (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Lewis B. Silverman, M.D., Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-001
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia in children; High Risk ALL; Standard Risk ALL; E. coli asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisone; Dexamethasone; Doxorubicin; Dexrazoxane; Vincristine; Methotrexate; Leucovorin; Asparaginase; Cytarabine; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Individualized ASP dose (Experimental)
  Interventions: Drug: doxorubicin; Drug: E. coli asparaginase; Drug: vincristine; Drug: methotrexate; Drug: Leucovorin; Drug: cytarabine; Drug: Methotrexate/Hydrocortisone
- Fixed dose ASP (Active Comparator)
  Interventions: Drug: doxorubicin; Drug: E. coli asparaginase; Drug: vincristine; Drug: methotrexate; Drug: Leucovorin; Drug: cytarabine; Drug: Methotrexate/Hydrocortisone
- Dexamethasone (Experimental)
  Interventions: Drug: dexamethasone; Drug: doxorubicin; Drug: vincristine; Drug: methotrexate; Drug: Leucovorin; Drug: Asparaginase; Drug: cytarabine; Drug: Methotrexate/Hydrocortisone
- Prednisone (Active Comparator)
  Interventions: Drug: prednisone; Drug: doxorubicin; Drug: vincristine; Drug: methotrexate; Drug: Leucovorin; Drug: Asparaginase; Drug: cytarabine; Drug: Methotrexate/Hydrocortisone

INTERVENTIONS:
Drug: prednisone — Induction Phase: Given orally or intravenously Days 0-28 Intensification Phase: Given orally Days 1-5 of each cycle Continuation Phase: Given orally Days 1-5 of each cycle
  Arms: Prednisone
Drug: dexamethasone — Intensification Phase: Given orally days 1-5 of each cycle Continuation Phase: Given orally days 1-5 pf each cycle
  Arms: Dexamethasone
Drug: doxorubicin — Induction Phase: Intravenously on Days 0,1 Intensification Phase: Intravenously on Day 1 of each cycle
  Other Names: dexrazoxane
Drug: E. coli asparaginase — Intensification Phase: In the muscle weekly. Dose will vary
  Arms: Fixed dose ASP; Individualized ASP dose
Drug: vincristine — Induction: Intravenously on days 0, 7, 14, 21 MLL Intensification Phase: Intravenously on Days 1, 8, 15, 22 CNS Therapy: Intravenously on Day 1 Intensification Phase: Intravenously on day 1 of each cycle Continuation Phase: Intravenously on Day 1 of each cycle
Drug: methotrexate — Induction: Intravenously on Day 2 MLL Intensification: Intravenously on Days 1, 8 Intensification: (when doxorubicin completed) Intravenously or into the muscle weekly Continuation: Intravenously or into the muscle weekly
Drug: Leucovorin — Induction Phase: Intravenously or orally begins 36 hours after methotrexate MLL Intensification: Intravenously or orally begins 36 hours after methotrexate
Drug: Asparaginase — Induction: Into the muscle on Day 4 MLL Intensification: Into the muscle on Days 16, 23
  Arms: Dexamethasone; Prednisone
Drug: cytarabine — Induction: Intrathecal on Days 0, 14, 28 MLL Intensification: Intravenously on Days 15, 16, 22, 23
  Other Names: ARA-C
Drug: Methotrexate/Hydrocortisone — Induction: Intrathecal on Days 14, 28 MLL Intensification: Intrathecal on Days 2,9

SUMMARY:
The purpose of this study is to reduce the side-effects from anti-leukemia therapy. The therapy in this study is based upon treatment information learned from prior clinical research programs as well as from laboratory research.

DETAILED DESCRIPTION:
* Children with acute lymphoblastic leukemia are treated somewhat differently depending on the relative risk of the leukemia recurring. Patients will be separated into "Standard Risk" and "High Risk".
* The treatment program for both groups is separated into 4 phases. The phases of treatment are induction, central nervous system (CNS) therapy, intensification and continuation.
* The induction phase of therapy lasts for about one month and its purpose is to kill all detectable leukemia cells. Patients in both groups will receive the following medication: prednisone, vincristine, doxorubicin, methotrexate, leucovorin, asparaginase, cytarabine (ARA-C), and hydrocortisone. Patients in the "Hight Risk" group will also receive dexrazoxane.
* Patients whose leukemia is found to have a specific genetic abnormality involving a gene on chromosome 11 (known as MLL gene) will have a MLL intensification phase which begins after complete remission and lasts about 1 month. The drugs involved in MLL intensification are: vincristine, methotrexate, leucovorin, hydrocortisone, cytarabine and L-asparaginase.
* CNS therapy begins immediately after the end of induction therapy, after remission is documented. This phase of treatment should last 3 weeks and includes a series of spinal taps with the instillation of anti-leukemia drugs. Four spinal taps will be performed over a two-week period. Both groups will receive vincristine, 6-mercaptopurine and methotrexate/cytarabine/hydrocortisone. Patients in the "High Risk" group will also receive doxorubicin with dexrazoxane.
* Radiation therapy will also be delivered to patients in the "High Risk" group during the CNS therapy phase. Radiation will be given in 8 daily treatments. The total dose of radiation used during this study is lower than what has been used in the past to help reduce side effects without increasing the risk of relapse.
* The intensification phase begins after the CNS therapy ends and lasts for 30 weeks. This phase is intended to further reduce the number of leukemia cells in the body and consists of cycles of chemotherapy repeated every three weeks with weekly shots of asparaginase. The drugs administered to both groups during this phase are: prednisone or dexamethasone, vincristine,6-mercaptopurine, methotrexate, E. coli asparaginase and cytarabine. Patients in the "High Risk" group will also receive doxorubicin and dexrazoxane.
* The continuation phase begins after the completion of the intensification phase and the goal is to eradicate all leukemia from the body. It consists of cycles of chemotherapy repeated every 3 weeks and is continued until the patient has been in remission for 2 years. The drugs administered during this phase are vincristine, prednisone or dexamethasone, 6-mercaptopurine, methotrexate and cytarabine.
* During this trial there are two randomizations, each is between the "standard" treatment and the "investigational" treatment. One randomization involves the drug E. coli L-asparaginase and two ways of dosing this drug. One way is to give the same standard dose of the drug that has been administered for years. The other way is to start with a lower dose and measure the amount of the drug in the blood every 3 weeks adjusting the dose as necessary. The goal of doing this is to maintain adequate drug levels with lower doses in the hope the it may reduce some side effects of the drug.
* The second randomization involves the drugs prednisone and dexamethasone. Both drugs have been used in the past to help treat ALL but it is not known if there is a difference between the two drugs, especially in terms of side effects. Patients will be randomized to either receive dexamethasone or prednisone.
* Throughout the study blood tests, urine tests, spinal taps, and bone marrow tests will be performed to monitor the disease status, side effects from medications and other complications from therapy.
* Quality of life questionnaires will also be performed by the patient (if older than 8), parent and patient's clinician.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia excluding known mature B-cell ALL by the presence of any of the following: surface immunoglobulin, L3 morphology, t(8;14) (q24;q32), t(8;22) or t(2;8)
* Age > 12 months but less than 18 years

Exclusion Criteria:

* Prior therapy except, 1 week of steroids, or emergent radiation therapy to the mediastinum
* Known HIV positive

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 498 (Actual)
Dates: Start 2000-09; Primary Completion 2004-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To optimize dosing of E. coli L-asparaginase during the intensification period | 5 years
To determine the side effects of prednisone versus dexamethasone. | 5 years

SECONDARY OUTCOMES:
To compare randomized treatment groups using health-related, quality-of-life analysis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Silverman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Background] Silverman LB, Gelber RD, Dalton VK, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Arkin S, Declerck L, Cohen HJ, Sallan SE. Improved outcome for children with acute lymphoblastic leukemia: results of Dana-Farber Consortium Protocol 91-01. Blood. 2001 Mar 1;97(5):1211-8. doi: 10.1182/blood.v97.5.1211. PMID 11222362
- [Background] Silverman LB, Declerck L, Gelber RD, Dalton VK, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Lipton JM, Cohen HJ, Sallan SE. Results of Dana-Farber Cancer Institute Consortium protocols for children with newly diagnosed acute lymphoblastic leukemia (1981-1995). Leukemia. 2000 Dec;14(12):2247-56. doi: 10.1038/sj.leu.2401980. PMID 11187916
- [Background] Goldberg JM, Silverman LB, Levy DE, Dalton VK, Gelber RD, Lehmann L, Cohen HJ, Sallan SE, Asselin BL. Childhood T-cell acute lymphoblastic leukemia: the Dana-Farber Cancer Institute acute lymphoblastic leukemia consortium experience. J Clin Oncol. 2003 Oct 1;21(19):3616-22. doi: 10.1200/JCO.2003.10.116. PMID 14512392
- [Background] Lipshultz SE, Rifai N, Dalton VM, Levy DE, Silverman LB, Lipsitz SR, Colan SD, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Gelber RD, Sallan SE. The effect of dexrazoxane on myocardial injury in doxorubicin-treated children with acute lymphoblastic leukemia. N Engl J Med. 2004 Jul 8;351(2):145-53. doi: 10.1056/NEJMoa035153. PMID 15247354
- [Derived] Vrooman LM, Stevenson KE, Supko JG, O'Brien J, Dahlberg SE, Asselin BL, Athale UH, Clavell LA, Kelly KM, Kutok JL, Laverdiere C, Lipshultz SE, Michon B, Schorin M, Relling MV, Cohen HJ, Neuberg DS, Sallan SE, Silverman LB. Postinduction dexamethasone and individualized dosing of Escherichia Coli L-asparaginase each improve outcome of children and adolescents with newly diagnosed acute lymphoblastic leukemia: results from a randomized study--Dana-Farber Cancer Institute ALL Consortium Protocol 00-01. J Clin Oncol. 2013 Mar 20;31(9):1202-10. doi: 10.1200/JCO.2012.43.2070. Epub 2013 Jan 28. PMID 23358966